CLINICAL TRIAL: NCT05418192
Title: Effects of Therapeutic Dosing Through Enriched Environment on Gross Motor Function and Spasticity in Spastic Quadriplegic Cerebral Palsy
Brief Title: Effects of Dosing and Environment on Gross Motor and Spasticity in Spastic Quadriplegic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC-UOL-/74-03/2022
Record Dates: First submitted 2022-06-08; First posted 2022-06-14 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Spastic Cerebral Palsy
Keywords: Therapeutic Dosing; Enriched Environment
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Intervention Given: Enriched Environment (age-appropriate) + NDT + Therapeutic Dosing
  Interventions: Other: Enriched Environment
- Group B (Other): Traditional Physical Therapy consisting of NDT
  Interventions: Other: Traditional Physcial Therapy

INTERVENTIONS:
Other: Enriched Environment — Enriched Environment (EE) consisted of motor and sensory enriched play environment to promote participant's self-generated movements, exploration and task success. EE also included positioning in a graded manner. Visual stimulus and level appropriate vestibular stimulus was also given. Dosing of positioning and sensory inputs was done throughout the therapy. Primary Intervention will be given for 20 to 25 minutes intermittently for period of 4-5 hours a day, 5 days a week for 24 weeks.
  Arms: Group A
Other: Traditional Physcial Therapy — Participants of this group received traditional physical therapy based NDT. No additional dosing guidance was given to this group. No home program was specifically assigned to this group. No specific environmental modifications were made for this group.
  Arms: Group B

SUMMARY:
This study focuses on how enriched environment along with the traditional physical therapy improves the gross motor function in spastic quadriplegic cerebral palsy children. And how much dosing is required to gain that clinically significant improvement.

DETAILED DESCRIPTION:
There is still a blurred area regarding dosage parameter in cerebral palsy rehabilitation. This study is focused primarily on the fact that level appropriate selection of time, type, frequency, and intensity of intervention (sensory and motor) plays a very vital role in developing gross motor functions. Secondly it is very important to establish the impact of enriched environmental inputs and foster parent capacity as an early intervention taking into account cerebral palsy (CP) specific positioning and handling along with level appropriate sensory inputs.

ELIGIBILITY:
Inclusion Criteria:

Age Group between 7 months to 5 years.

* Spastic Quadriplegia
* Gross Motor Function Classification System (GMFCS) level IV and V
* Modified Ashworth Scale (MAS): level 2
* Both Gender

Exclusion Criteria:

* History of fits

  * Medications
  * Dislocation and fracture
  * Visual/Auditory Impairment
  * Patients taking therapy from multiple places

Ages: 7 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 82 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Gross Motor Function | 5 months
  To check the improvement in gross motor function on Gross Motor Functional Measure scale of spastic quadriplegic cerebral palsy children. The scoring system of this scale is divided into five dimensions of gross motor function:(a) lying and rolling, (b) sitting, (c) crawling and kneeling, (d) standing, and (e) walking, running and jumping. The scoring is done on four points: 0=does not initiate
  1. = initiates
  2. = partially completes
  3. = completes Higher scores mean better outcome whereas low scores show little to no improvement in gross motor function.

SECONDARY OUTCOMES:
Spasticity | 5 months
  To check the improvement in spasticity on Modified Ashworth Scale scale in spastic quadriplegic cerebral palsy children. The Modified Ashworth Scale is a 6-point scale. Scores range from 0 to 4, where lower scores represent normal muscle tone and higher scores represent spasticity or increased resistance to passive movement.

CONTACTS AND LOCATIONS:
Overall Officials: Safa Saleem, DPT, Principal Investigator — University of Lahore
Locations (1):
- The University of Lahore Teaching Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No